CLINICAL TRIAL: NCT02726334
Title: A Phase I, Dose Escalation Study of BNC101 (Anti-LGR5 Humanized Monoclonal Antibody) in Patients With Metastatic Colorectal Cancer.
Brief Title: A Phase I, Dose Escalation Study of BNC101 in Patients With Metastatic Colorectal Cancer.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Monotherapy arm completed. Combination arm did not proceed (sponsor decision).
Sponsor: Bionomics Limited (Industry)
Collaborators: CPR Pharma Services Pty Ltd, Australia (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BNC101. 001
Record Dates: First submitted 2016-03-28; First posted 2016-04-01 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Colorectal Cancer
Keywords: Metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group/Stream 1 - Monotherapy (Experimental): Patient group: Patients who have failed at least two lines of chemotherapy for metastatic disease.
  Treatment: BNC101 administered via intravenous infusion over 60 minutes weekly.
  Patients with stable disease or a response at or after day 56 (2 cycles) will be allowed to continue to receive weekly doses of BNC101 until disease progression.
  Interventions: Drug: BNC101 Solution for Infusion
- Group/Stream 2 - Combination Chemo (Experimental): Patient Group: Patients who have failed at least one line of chemotherapy for metastatic disease.
  Treatment: BNC101 administered in combination with FOLFIRI
  Participants will be treated until disease progression, intolerable toxicity, withdrawal of consent, or study termination by the Sponsor, whichever occurs first.
  Interventions: Drug: BNC101 in combination with FOLFIRI

INTERVENTIONS:
Drug: BNC101 Solution for Infusion — Administration: Administered via IV infusion once a week over 60 minutes (1 hour).
  Other Names: BNC101
  Arms: Group/Stream 1 - Monotherapy
Drug: BNC101 in combination with FOLFIRI — BNC101 - Starting dose as determined by Arm A portion (one dose level below recommended Phase 2 dose).
  BNC101 Administration: Administered via IV Infusion once a week over 60 minutes (1 hour).
  FOLFIRI components:
  Irinotecan (IRI) - Starting dose 180 mg/m2 (over 90 minutes on Day 1) Leucovorin (LV) - Starting dose 400 mg/m2 (administered over 120 minutes on Day 1 concurrently with IRI) 5-FU bolus - Starting dose 400 mg/m2 (administered after LV on Day 1, then) 5-FU infusion - Starting dose 2400 mg/m2 (administered over 48 hours starting on Day 1)
  FOLFIRI Cycles are repeated every 14 days.
  Other Names: FOLFIRI
  Arms: Group/Stream 2 - Combination Chemo

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (which will be the dose recommended for a Phase 2 study), safety, tolerability and pharmacokinetic profile (study of movement of the drug within the body, including absorption and distribution) of the study drug, BNC101 when administered intravenously as a single agent or in combination with chemotherapy in patients with metastatic colorectal cancer who have failed at least 1 or 2 lines of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written Informed Consent
2. Age > 18 years
3. Eastern Cooperative Oncology Group (ECOG) score 0 - 1.
4. Histologically or cytologically confirmed colorectal cancer patients who have failed at least 2 lines of chemotherapy (monotherapy treatment cohorts) or at least 1 line of chemotherapy (combination treatment cohorts) for metastatic disease, and in the opinion of both physician and patient it is not unreasonable to try experimental therapy. Adjuvant FOLFOX within the last 6 months is considered a line of therapy. A maintenance strategy post 1st line treatment is not considered as an additional line of therapy.
5. Patients must have accessible tumor lesions amenable to biopsy which would not put the patient or their treatment at risk. Patients in monotherapy escalation cohort 3 and onwards, the monotherapy expansion cohort, and all combination treatment patients, agree and are willing to provide 2 serial tumor lesion biopsies (a minimum of 2 fresh cores/punches preferred whenever possible). Biopsies can be from liver metastases, in lieu of the primary tumor. The presence of tumor tissue in fresh biopsies is to be certified by a trained pathologist using appropriate extemporaneous histology or cytology procedures. Refer to Appendix 6 for biopsy procedures.
6. All AEs of any prior chemotherapy, surgery, or radiotherapy, must have resolved to Grade ≤ 1.
7. Measurable or evaluable disease per RECIST version 1.1.
8. No known brain metastases (see also exclusion criterion No. 10).
9. Life expectancy of at least > 12 weeks.
10. Normal organ and marrow function:

    1. Absolute neutrophil count (ANC) > 1,500/mL without growth factor support in the past 14 days prior to enrolment
    2. Platelets > 100,000/mL without transfusions in the past 14 days prior to enrolment
    3. Hemoglobin > 9.0 g/dL - Patients may be transfused or receive erythropoietic treatment to meet this criterion
    4. Total bilirubin < 1.5 x institutional upper limit of normal (ULN) (< 2 x ULN for subjects with Gilbert's syndrome)
    5. Serum albumin ≥ 3 g/dL.
11. Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase, SGOT) and alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase, SGPT) < 2.5 x institutional ULN (for subjects with hepatic involvement < 5 x institutional ULN but cannot be associated with elevated bilirubin).
12. Alkaline phosphatase (AlkPhos) > 2.5 x ULN, except in patients with documented liver or bone metastases, where it can be < 5 x ULN.
13. For patients receiving biopsies, prothrombin time (PT) and activated partial thromboplastin time (APTT)/international normalized ratio (INR) within normal limits (± 15%)..
14. Creatinine < 1.5 x institutional ULN OR Creatinine clearance > 60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal based on the Cockroft-Gault glomerular filtration rate estimation:

(140 - age) x (weight in kg) x (0.85 if female)

72 x (serum creatinine in mg/dL)

(NOTE: For patients with a Body Mass Index (BMI) > 30 kg/m2, lean body weight should be used instead)

15. No clinically significant abnormalities in urinalysis results (obtained ≤ 14 days prior to enrolment).

16. No current or recent (within 3 months of study drug administration) gastrointestinal disease such as chronic or intermittent diarrhea, or disorders that increase the risk of diarrhea, such as inflammatory bowel disease. Non-chronic conditions (e.g., infectious diarrhea) that are completely resolved for at least 2 weeks prior to starting study treatment is allowed.

17. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form of contraception (e.g., surgical sterilization, a reliable barrier method, birth control pills, or contraceptive hormone implants) and to continue its use for 6 months after the last dose of study drugs.

18. Women of childbearing potential must have a negative serum pregnancy test (β-hCG) within 72 hours prior to first study drug administration.

Exclusion Criteria:

1. Inability to comply with study and follow-up procedures (including, but not limited to: geographical or administrative reasons, and planned vacation absences for more than 7 consecutive days during the study).
2. Women who are pregnant or lactating.
3. Colorectal cancer patients going on to receive 1st line therapy for metastatic disease.
4. Treatment with chemotherapy, immunotherapy, biologic therapy, or radiation therapy as cancer therapy within 4 weeks before initiation of study treatment. Six weeks should have elapsed if prior chemotherapy treatment included nitrosoureas or mitomycin C.
5. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to Day 1 of Cycle 1.
6. Patients who have received antibody-based therapies within 28 days or 5 half-lives of the agent, whichever is longer.
7. Major surgery, other than diagnostic surgery, within 6 weeks before first study drug administration.
8. Clinically detectable (by physical exam) third-space fluid collections (e.g., ascites or pleural effusion) that cannot be controlled by drainage or other procedures prior to study entry.
9. Any uncontrolled medical or psychiatric risk factors which would contraindicate the use or impair the ability of the patient to provide informed consent, receive protocol therapy or may impose excessive risk to the patient.
10. Central nervous system (CNS) metastases, unless previously treated and well-controlled for at least 3 months (defined as clinically stable, no edema, no steroids and stable in 2 scans at least 4 weeks apart). Patients who display signs or symptoms of CNS metastases or should be imaged with CT or magnetic resonance imaging (MRI) of the head. Should metastases, including meningeal deposits be detected, these patients will not be treated with BNC101.
11. Current use of medications that may have the potential of QTc prolongation (refer to Appendix 1). If the need for use of these medications arises during the study, a discussion with and approval by the sponsor would be required.
12. History of allergy or hypersensitivity to Chinese Hamster Ovary cell products, any compound of the BNC101 formulation, or any of the chemotherapy agents to be used in this study.
13. Active uncontrolled bacterial, viral, or fungal infection, requiring systemic therapy.
14. Patient has known infection with human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C, alcoholic or other hepatitis, or cirrhosis.
15. Inability to be venipunctured and/or tolerate venous access.
16. Second malignancies within 5 years prior to enrolment, except for those with a negligible risk of metastasis or death, such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent.
17. Active autoimmune disease that is not controlled by nonsteroidal anti-inflammatory drugs, inhaled corticosteroids, or the equivalent of > 10 mg/day prednisone.
18. Seizure disease requiring current anticonvulsant treatment.
19. History of inflammatory bowel disease (active or past) or active peptic ulcer disease.
20. History of chronic leukemias (e.g., chronic lymphocytic leukemia).
21. History of previous, whole abdomen radiation therapy (or total pelvic radiation therapy in rectal cancer patients) or more than Grade 1 residual toxicity from previous radiation therapy. NOTE: Patients with previous standard, routine abdomino-pelvic radiotherapy are eligible and not encompassed by this criterion, which only applies to whole abdomen or total pelvic radiotherapy.
22. Patients with high cardiovascular risk, including, but not limited to coronary stenting in the previous 3 months or myocardial infarction in the past year [Patients with New York Heart Association (NYHA) class I classification are acceptable].
23. Congenital or acquired long QT syndrome.
24. QTc prolongation defined as a QTc interval greater than or equal to 450 msec at baseline; interval determination will be based on a mean value obtained from 3 baseline ECGs obtained at least 5 minutes apart.
25. Patients with history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | DLT period of 28 days per dose level
  To determine the maximum tolerated dose (MTD) of BNC101, both as single agent and in combination chemotherapy in metastatic colorectal cancer patients.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria